CLINICAL TRIAL: NCT02273479
Title: Pharmacokinetics and Safety of Asasantin Extended Release (RAD-SP) 200/25 mg Capsules b.i.d. in Randomised, Double-blind, Placebo-controlled Study in Japanese Healthy Male Volunteers
Brief Title: Pharmacokinetics and Safety of Asasantin Extended Release (RAD-SP) Capsules in Japanese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9.127
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin, Dipyridamole Drug Combination

ARMS (2):
- Asasantin® (Experimental)
  Interventions: Drug: Asasantin®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asasantin® — Asasantin® extended release (RAD-SP)
  Arms: Asasantin®
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate pharmacokinetics, pharmacodynamics and safety of RAD-SP capsule in multiple administration to healthy adult male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers judged by the investigator as appropriate subjects on the basis of screening test results
* Age range: ≥ 20 years and ≤ 35 years
* Body weight between 50 and 80 kg
* Obesity is within ± 20% of the standard body weight
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* History of drug allergy
* History of bronchial asthma
* History of drug abuse and alcohol abuse
* History of hemorrhagic tendency or hemorrhagic disease
* Volunteers who have experiences in playing sports such as boxing which may damage the brain
* Accidents associated with brain concussion and contusion (traffic accident, etc.)
* Administration of other study drug within 4 months before start of administration of this study drug
* Collection of whole blood (≥ 400 ml) within 3 months before study drug administration
* Collection of component blood (≥ 400 ml) within 1 months before study drug administration
* Intake of some drug or other within 10 days before the study drug administration
* Excessive physical activities within the last 5 days prior to study drug administration
* Intake of alcohol within 3 days before study drug administration
* Volunteers judged by the investigator to be inappropriate as the subjects of study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 1999-07; Primary Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve at steady state (AUCss) | up to 144 hours after first drug administration
Maximum drug plasma concentration at steady state (Cmax,ss) | up to 144 hours after first drug administration
Cmax,ss/AUCss | up to 144 hours after first drug administration
Minimum drug plasma concentration at steady state (Cmin,ss) | up to 144 hours after first drug administration
Time to reach Cmax (tmax) | up to 144 hours after first drug administration
Terminal half-life (t1/2) | up to 144 hours after first drug administration
Mean residence time (MRT) | up to 144 hours after first drug administration
Percent peak trough fluctuation (%PTF) | up to 144 hours after first drug administration

SECONDARY OUTCOMES:
Platelet adenosine uptake inhibition rate (AUI) | up to 74 hours after first drug administration
Malondialdehyde (MDA) production inhibition rate | up to 74 hours after first drug administration
Thromboxane B2 (TXB2) production inhibition rate | up to 74 hours after first drug administration
Number of subjects with adverse events | up to 14 days after first drug administration
Number of subjects with abnormal changes in laboratory parameters | up to 14 days after first drug administration
Number of subjects with abnormal changes in vital signs | up to 14 days after first drug administration
Number of subjects with abnormal changes in electrocardiogram findings | up to 14 days after first drug administration